CLINICAL TRIAL: NCT04020822
Title: Feasibility Study of New Subcutaneous Glucose Sensor With Recording Devices - Phase 3 Group
Brief Title: Feasibility Study of New Subcutaneous Glucose Sensor With Recording Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP318
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: Acetaminophen
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Subjects Wearing Guardian Sensor (3)s (Experimental): Each subject will wear 4 Guardian Sensor (3)s connected to a Guardian Link (3) Transmitter and/or Guardian Connect Transmitter for 11 days of sensor wear.
  Interventions: Device: Guardian Sensor (3)

INTERVENTIONS:
Device: Guardian Sensor (3) — Guardian Sensor (3) connected to Guardian Link (3) Transmitter and/or Guardian Connect Transmitter.

SUMMARY:
The purpose of Phase 3 Group is to evaluate the impact of acetaminophen on the performance of Guardian Sensor (3) during 11 days of wear (approximately 264 hours) in subjects with insulin requiring diabetes,18-75 years of age.

DETAILED DESCRIPTION:
The study is a multi-center, prospective single-arm design without controls. All subjects will be assigned to treatment for 11 days of sensor wear. Each subject will wear 4 Guardian Sensor (3)s, and each will be connected to a Guardian Link (3) Transmitter and/or Guardian Connect Transmitter. Subjects will not use sensor glucose values for diabetes management.

On days 1, 3, 5, and 6, subjects will be asked to measure blood glucose (BG) using a home glucose meter approximately every 20 minutes for 5 hours. Subjects will be asked to take one gram of acetaminophen orally on days 3, 5, and 6 of sensor wear.

On day 11, devices will be removed, data uploaded from the study meter and transmitter or recorder, skin assessment will be performed, and the subject's participation in the study will be completed.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18-75 years of age at time of screening
2. A clinical diagnosis of type 1 or type 2 diabetes as determined by investigator, for at least the last 12 months
3. Subject is using insulin to treat their diabetes
4. Subject agrees to comply with the study protocol requirements
5. Subject is willing to perform self-monitoring of blood glucose approximately every 20 minutes during FST

Exclusion Criteria:

1. Subject has history of allergy to acetaminophen or has been told by health care provider they may not ingest acetaminophen
2. Subject reports history of liver cirrhosis or problems with liver that a health care provider told them they should not use acetaminophen because of liver disorder.
3. Subject is unable to tolerate tape adhesive in the area of sensor placement
4. Subject has any unresolved adverse skin condition in the area of sensor or device placement (e.g. psoriasis, rash, Staphylococcus infection)
5. Subject is actively participating in or plans to enroll in an investigational study (drug or device), other than this study, wherein they have received treatment from an investigational drug or device
6. Subject has a positive urine pregnancy test at time of screening
7. Subject is female, sexually active without the use of contraception, able to become pregnant or plans to become pregnant during the course of the study
8. Subject is unwilling to participate in study procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-08-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Barbara Davis Center for Diabetes, Aurora, Colorado
  - Atlanta Diabetes Associates, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subjects Wearing Guardian Sensor (3)s
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Subjects Wearing Guardian Sensor (3)s
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.9 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Sensor Glucose Before and After Acetaminophen Administration
Description: Accuracy (mean absolute relative difference) between the primary sensor values and meter BG values during the hour leading to and two hours after ingestion of acetaminophen. Primary sensor will be assigned to sensor number one (inserted in arm).
  Mean Absolute Relative Difference = Mean of ((absolute difference of meter and sensor blood glucose values / meter glucose values) * 100).
  Note that the results reported below for one hour leading to and two hours after acetaminophen ingestion were pooled together across multiple testing days (days 3, 5, and 6).
Time Frame: Assessed up to 11 days, frequent sample testing recordings from the three-hour period leading to and after Acetaminophen ingestion on days 3, 5, and 6 reported
Population: Only data from 13 subjects were evaluated due to data loss.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Subjects Wearing Guardian Sensor (3)s
Number analyzed (Participants) | 13
Percent
  (-1, 0] hour of Acetaminophen Ingestion | 9.46 (4.63)
  (0, 1] hour of Acetaminophen Ingestion | 12.02 (6.53)
  (1, 2] hour of Acetaminophen Ingestion | 16.98 (10.96)

ADVERSE EVENTS:
Time Frame: 11 Days
Arm/Group | Subjects Wearing Guardian Sensor (3)s
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/22/NCT04020822/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/22/NCT04020822/SAP_001.pdf